CLINICAL TRIAL: NCT06316271
Title: Endothelial Dysfunction and Cardiovascular Remodeling in Pathophyisiology of Prehypertension
Brief Title: Endothelial Function in Prehypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: University Hospital Center Osijek (Unknown)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science Faculty of Medicine Osijek, Josip Juraj Strossmayer University of Osijek
Other Study IDs: PreHT 2024
Record Dates: First submitted 2024-03-02; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Hypertension,Essential
Keywords: hypertension; prehypertension; endothelium; left ventricle; hemodynamics
MeSH Terms: conditions — Essential Hypertension; Hypertension; Prehypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, peripheral blood mononuclear cells (PBMCs)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normotensive Group: BP less than or equal to 129/84 mmHg
- Prehypertensive Group: BP 130-139/85-89 mmHg
- Hypertensive Group: BP 140-150/90-100 mmHg

SUMMARY:
In the frame of this proposal investigators will test the hypothesis that high normal blood pressure (prehypertension; PreHT) induces systemic endothelial dysfunction and endothelial activation in both micro- and macrocirculation, reduces re-endothelialization potential of human endothelial progenitor cells (EPCs) and increases the level of endothelial extracellular vesicles (EVs), which are accompanied by increased oxidative stress level. Furthermore, initial vascular and left ventricle (LV) remodeling contributes to changes in systemic hemodynamics and may be influenced by altered regulatory role of renin-angiotensin system (RAS) and autonomic nervous system (ANS) in PreHT but otherwise healthy individuals. To distinguish high normal blood pressure effect from those considered normal or high, study will be performed in three groups of individuals: prehypertensive (BP 130-139/85-89 mmHg), hypertensive (stage I, BP 140-150/90-100 mmHg), and controls (BP less than or equal to 129/85 mmHg). Altogether, the impairment of normal vascular relaxation mechanisms, endothelial activation as well as vascular and LV remodeling could play crucial role in increased cardiovascular risk and CVDs incidence in PreHT individuals. Moreover, the prognostic significance of assessing endotehlial dysfunction in hypertension (as well as in PreHT) is yet to be established.

ELIGIBILITY:
Inclusion Criteria:

* adults of both sexes with normotensive, prehypertensive and grade I hypertension blood pressure values

Exclusion Criteria:

* cardiovascular diseases, but grade I hypertension (BP 140-150/90-100 mmHg)
* diabetes
* kidney disease
* cerebrovascular diseases
* peripheral artery disease
* taking oral contraceptives or any drugs that could affect the endothelium

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects will be divided in the three study groups based on BP assessment using ambulatory blood pressure monitoring (ABPM). Hypertensive group will include only newly diagnosed patients who have not taken antihypertensive therapy.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic microvascular function | Day 1
  Skin microvascular reactivity assessed by Laser Doppler flowmetry (post-occlusive reactive hyperemia, iontophoresis of acetylcholine and sodium nitroprusside, local thermal hyperemia) - measured in perfusion units (PU)
Systemic macrovascular function | Day 1
  Vascular ultrasound measurement of brachial artery flow mediated dilation (FMD)
Aortic stiffness | Day 1
  Measurement of pulse wave velocity (PWV) using impedance cardiography.
Left ventricle global longitudinal strain | Day 1
  Global longitudinal strain (GLS) of left ventricle obtained by two-dimensional speckle tracking echocardiography.

SECONDARY OUTCOMES:
Oxidative stress - 8-iso-prostaglandin F2α (8-iso-PGF2α) | Day 1
  ELISA measurement of serum 8-iso-PGF2α concentration. 8-iso-PGF2α is an isoprostane that is produced by the non-enzymatic peroxidation of arachidonic acid in membrane phospholipids.
Activity of renin-angiotensin system (RAS) | Day 1
  ELISA measurement of plasma renin activity (PRA).
Endothelial progenitor cells (EPCs) | Day 1
  Detection of EPCs using a two laser flow cytometer (FacsCanto II, Becton Dickinson) and CBA kits (cytometry beads assays).
Endothelial extracellular vesicles (eEVs) | Day 1
  Detection of eEVs using a two laser flow cytometer (FacsCanto II, Becton Dickinson) and CBA kits (cytometry beads assays).
Systemic peripheral vascular resistance | Day 1
  Systemic peripheral vascular resistance assessement using non-invasive impedance cardiography (ICG).
Autonomic nervous system (ANS) activity | Day 1
  Assessment of a 5-minute heart rate variability (5-min HRV).
Matrix metalloproteinase 9 | Day 1
  ELISA measurement of serum matrix metalloproteinase 9 level.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No